CLINICAL TRIAL: NCT01460654
Title: Testosterone and Alendronate in Hypogonadal Men
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Endo Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGH-988
Record Dates: First submitted 2011-10-20; First posted 2011-10-27 (Estimated); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hypogonadism; Osteopenia; Osteoporosis
MeSH Terms: conditions — Hypogonadism; Bone Diseases, Metabolic; Osteoporosis | interventions — Testosterone; Alendronate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Testosterone and Placebo Alendronate (Placebo Comparator)
  Interventions: Drug: Testosterone; Drug: Placebo Alendronate
- Alendronate and Placebo Testosterone (Placebo Comparator)
  Interventions: Drug: Alendronate; Drug: Placebo Testosterone
- Testosterone and Alendronate (Experimental)
  Interventions: Drug: Testosterone; Drug: Alendronate

INTERVENTIONS:
Drug: Testosterone — Testosterone Gel (Fortesta) 40mg daily.
  Arms: Testosterone and Alendronate; Testosterone and Placebo Alendronate
Drug: Alendronate — Alendronate (Fosamax) 70mg every week.
  Arms: Alendronate and Placebo Testosterone; Testosterone and Alendronate
Drug: Placebo Alendronate — A placebo alendronate tablet will be taken every week by subjects in the Testosterone and Placebo Alendronate Group.
  Arms: Testosterone and Placebo Alendronate
Drug: Placebo Testosterone — Placebo testosterone gel will be applied daily by subjects in the Alendronate and Placebo Testosterone group.
  Arms: Alendronate and Placebo Testosterone

SUMMARY:
This study will investigate the hypothesis that the combination of testosterone replacement and alendronate will improve bone density and parameters of bone quality more than either medication alone in older men with low testosterone levels and low bone density.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 60 or above
* Testosterone <300 ng/dL
* DXA T score < -1 OR FRAX Score of 3% or greater for hip fracture or 20% or greater for major osteoporotic fracture

Exclusion Criteria:

* Significant liver or kidney disease
* Elevated prolactin level
* Abnormal TSH
* Abnormal 25-Vitamin D
* PSA > 2.5
* History of malignancy
* Calcium > 10.6
* Alkaline Phosphatase > 150
* Fracture within the last 6 months
* History of acute urinary retention
* Hematocrit < 32% or > 50%
* Fracture within the past 6 months
* American Urological Association BPH symptom index > 21
* Sleep apnea
* Abnormalities of the esophagus which delay esophageal emptying
* Significant cardiopulmonary disease

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone and Placebo Alendronate | Alendronate and Placebo Testosterone | Testosterone and Alendronate
Started | 19 | 10 | 15
Completed | 14 | 9 | 13
Not Completed | 5 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone and Placebo Alendronate | Alendronate and Placebo Testosterone | Testosterone and Alendronate | Total
Number analyzed (Participants) | 19 | 10 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 7
  >=65 years | 17 | 8 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (4.9) | 70.1 (6.5) | 69.8 (5.1) | 69.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 19 | 10 | 15 | 44
Region of Enrollment [Number; unit: participants]
  United States | 19 | 10 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Spine Bone Density From Baseline to 12 Months
Description: Percent Change in Spine Bone Density from Baseline (month 0) to Month 12
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent change of bone mineral density
Arm/Group | Testosterone and Placebo Alendronate | Alendronate and Placebo Testosterone | Testosterone and Alendronate
Number analyzed (Participants) | 14 | 9 | 13
percent change of bone mineral density | 2.52 (0.02) | 0.61 (0.03) | 3.16 (0.04)

ADVERSE EVENTS:
Arm/Group | Testosterone and Placebo Alendronate | Alendronate and Placebo Testosterone | Testosterone and Alendronate
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/10 | 0/15
Other Adverse Events (participants affected / at risk) | 13/19 | 8/10 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone and Placebo Alendronate (N=19) | Alendronate and Placebo Testosterone (N=10) | Testosterone and Alendronate (N=15)
nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
bladder cancer (Renal and urinary disorders) | 1 | 0 | 0
spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone and Placebo Alendronate (N=19) | Alendronate and Placebo Testosterone (N=10) | Testosterone and Alendronate (N=15)
chest discomfort (Cardiac disorders) | 3 | 0 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
dizziness (Nervous system disorders) | 1 | 0 | 1
hypertension (Cardiac disorders) | 1 | 1 | 0
glaucoma (Eye disorders) | 1 | 0 | 0
Shingles (Infections and infestations) | 1 | 0 | 0
Sinus surgery (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
hypoglycemia (Endocrine disorders) | 0 | 1 | 1
Elevated hematocrit (Blood and lymphatic system disorders) | 0 | 2 | 0
Sciatic nerve pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
prostate nodule (Renal and urinary disorders) | 0 | 1 | 0
hematuria (Renal and urinary disorders) | 0 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 0 | 1
Elevated creatinine (Renal and urinary disorders) | 0 | 0 | 1
Elevated prostrate screen antigen (Renal and urinary disorders) | 0 | 0 | 1
Crohns disease (Gastrointestinal disorders) | 0 | 0 | 1
plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
muscle ache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
achilles tendon tear (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No